CLINICAL TRIAL: NCT01648933
Title: Perfusion Analysis Using Rubidium in Cardiac Sarcoidosis
Acronym: PARCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOR10027
Record Dates: First submitted 2012-04-12; First posted 2012-07-25 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; heart; Rubidium; PET
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sarcoidosis (Experimental): Rubidium PET:
  Myocardial Perfusion Imaging
  Interventions: Radiation: Rubidium PET

INTERVENTIONS:
Radiation: Rubidium PET — Myocardial Perfusion Imaging

SUMMARY:
The study aims at assessing diagnostic and therapeutic impact of Rubidium-82 PET in cardiac sarcoidosis.

DETAILED DESCRIPTION:
The presence of cardiac involvement is a serious complication of sarcoidosis. Early diagnosis is challenging since it relies on an array of clinical, biological and imaging abnormalities. Myocardial perfusion imaging with sestamibi is currently a major feature of the diagnosis, since it allows to evidence both microcirculatory impairments and scar. However, some technical limitations are inherent to SPECT, mainly poor spatial resolution and lack of attenuation correction, resulting in the absence of flow quantification. Rubidium-82 (Rb) PET proved to be more sensitive and specific than sestamibi SPECT in the diagnosis of coronary artery disease. Furthermore, it allows noninvasive measurement of coronary flow reserve. Finally, it exposes patients to lower radiation dose than SPECT. Therefore, Rb PET may help to better identify cardiac involvement of sarcoidosis, and hence to better select those patients who require high-dose steroids.

ELIGIBILITY:
Inclusion Criteria:

* (1) histologically proven sarcoidosis;
* (2) suspicion of cardiac involvement on symptoms, and/or ECG and/or echocardiogram.

Exclusion Criteria:

* patient < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
percentage of patient who has two different diagnostic and therapeutic attitude before knowing Rubidium-82 PET result and after knowing Rubidium-82 PET result | 60 days
  to assess diagnostic and therapeutic impacts of myocardial perfusion analysis with Rubidium-82 PET in cardiac sarcoidosis.

SECONDARY OUTCOMES:
Analysis of the cost for the use of Sestamibi SPECT and Rb-PET as MPI agents in cardiac sarcoidosis. | 9 months
  to compare the cost between the two exams and the health-economic impact of Sestamibi SPECT and Rb-PET as MPI agents in cardiac sarcoidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Le Guludec, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard 46, rue Henri-Huchard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided